CLINICAL TRIAL: NCT03528226
Title: Impact of Exercise Training on Endothelial Function in Adults With Type 1 Diabetes
Brief Title: Exercise Training and Endothelial Function in Type 1 Diabetes
Acronym: EVaDia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016_45.1; 2017-A02873-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-05-03; First posted 2018-05-17 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type1diabetes
Keywords: Type 1 diabetes; endothelial function; exercise training; physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training (Experimental)
  Interventions: Behavioral: Exercise Training Procedure
- Control (Other)
  Interventions: Behavioral: Normal life procedure

INTERVENTIONS:
Behavioral: Exercise Training Procedure — Exercise training: 3 sessions - 2 supervised and 1 unsupervised - per week of 30-60 min at 65% - 80% of maximum heart rate (4 months)
  Arms: Exercise Training
Behavioral: Normal life procedure — No supervised exercise training during the 4 month period.
  Arms: Control

SUMMARY:
Endothelial dysfunction and vasoreactivity disorders are early subclinical complications of type 1 diabetes (T1D). In a preventive setting, in T1D patients still free of complications, the research of non-pharmacological interventions to improve endothelial function appears fundamental.

In this randomized controlled trial, the effects of exercise training on endothelial function will be evaluated in T1D adults. Secondary objectives are to evaluate the exercise training effects on the micro and macrovascular function and exercise-induced tissue vasoreactivity and their possible neurometabolic consequences.

An improvement in vascular function, particularly endothelium-dependent, as well as in neurometabolic profile, through this non-pharmacological strategy is expected

ELIGIBILITY:
Inclusion Criteria:

* Covered by social security
* With a T1Diabete, diagnosed for at least 1 year, and free from macrovascular and microvascular diabetic complications.

Exclusion Criteria:

* type 1 diabetes diagnoses for less than 1 year
* MODY diabetes, mitochondrial diabetes or type 2 diabetes
* presence of macrovascular and/or microvascular diabetic complications (retinopathy, nephropathy, neuropathy ,…)
* Obesity (Body Mass Index > 30 kg/m²
* Smokers
* Hypertension
* Disabling painful discomfort for trunk, upper or lower limb movements
* Active chronic disease or in remission (excluding type 1 diabetes)
* Head trauma in the past

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in percent flow-mediated dilation (FMD) values | between baseline and at 4 months

SECONDARY OUTCOMES:
Change the vascular responses | at baseline , at 2 months , at 4 months
  Endothelium-dependent vasodilation capacity induced by post-occlusive reactive hyperaemia (5min occlusion) at the level of microcirculation (skin capillaries and arterioles of the hand)
  -Vasoreactivity of the cutaneous capillaries of the forearm in response to acetylcholine and sodium nitroprusside (iontophoresis)
Change the vascular responses | at baseline , at 2 months , at 4 months
  Endothelium-dependent vasodilation capacity induced by post-occlusive reactive hyperaemia (5min occlusion) at the level of microcirculation (skin capillaries and arterioles of the hand)
  -Dilatatory macrocirculation (brachial artery) and microcirculatory (capillaries of the hand) to nitroglycerine (in sublingual spraying)
Change the vascular responses | at baseline , at 2 months , at 4 months
  Endothelium-dependent vasodilation capacity induced by post-occlusive reactive hyperaemia (5min occlusion) at the level of microcirculation (skin capillaries and arterioles of the hand)
  -Evolution of the blood volume at the vastus lateralis muscle and the prefrontal cortex in response to an incremental maximal exercise
Change in percent flow-mediated dilation (FMD) values | between baseline and at 2 months
change the maximum oxygen consumption ( VO2max) | at baseline , at 2 months , at 4 months
Change Blood marker concentrations of nitric oxide (NO) | at baseline , at 2 months , at 4 months
change Blood concentration of neurotrophic factors | at baseline , at 2 months , at 4 months
  Blood concentration of neurotrophic factors and blood markers of metabolic profile
Body composition (DEXA) | at baseline , at 2 months , at 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Fontaine, MD,Phd, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France